CLINICAL TRIAL: NCT00982046
Title: A Clinical Comparison of Three Contact Lens Care Systems and Their Effect on Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: M-09-05
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2012-07

CONDITIONS: Contact Lenses
Keywords: contact lenses; disinfection solutions; contact lens care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ACUVUE OASYS (Active Comparator): Acuvue Oasys contact lenses worn on a daily wear basis and cleaned nightly with one of three contact lens care solutions. Each solution was used for 2 weeks, and the order in which the solutions were used was randomized. A fresh pair of lenses was dispensed with each solution. Total duration of contact lens wear was six weeks.
  Interventions: Device: Opti-Free RepleniSH multi-purpose disinfecting solution; Device: ReNu MultiPlus multi-purpose solution; Device: Clear Care cleaning and disinfecting system; Device: Senofilcon A contact lens (ACUVUE OASYS)
- AIR OPTIX AQUA (Active Comparator): Air Optix Aqua contact lenses worn on a daily wear basis and cleaned nightly with one of three contact lens care solutions. Each solution was used for 2 weeks, and the order in which the solutions were used was randomized. A fresh pair of lenses was dispensed with each solution. Total duration of contact lens wear was six weeks.
  Interventions: Device: Opti-Free RepleniSH multi-purpose disinfecting solution; Device: ReNu MultiPlus multi-purpose solution; Device: Clear Care cleaning and disinfecting system; Device: Lotrafilcon B contact lens (AIR OPTIX AQUA)
- Biofinity (Active Comparator): Biofinity contact lenses worn on a daily wear basis and cleaned nightly with one of three contact lens care solutions. Each solution was used for 2 weeks, and the order in which the solutions were used was randomized. A fresh pair of lenses was dispensed with each solution. Total duration of contact lens wear was six weeks.
  Interventions: Device: Opti-Free RepleniSH multi-purpose disinfecting solution; Device: ReNu MultiPlus multi-purpose solution; Device: Clear Care cleaning and disinfecting system; Device: Comfilcon A contact lens (Biofinity)

INTERVENTIONS:
Device: Opti-Free RepleniSH multi-purpose disinfecting solution — Contact lens solution CE-marked for intended use.
  Other Names: Opti-Free® RepleniSH®
Device: ReNu MultiPlus multi-purpose solution — Contact lens solution CE-marked for intended use.
  Other Names: ReNu® MultiPlus®
Device: Clear Care cleaning and disinfecting system — Contact lens care system CE-marked for intended use.
  Other Names: Clear Care®
Device: Senofilcon A contact lens (ACUVUE OASYS) — Silicone hydrogel contact lens worn for two weeks on a daily wear basis and cleaned nightly with one of three contact lens care solutions. The order of solutions was randomized, and a fresh pair of lenses was dispensed with each solution.
  Other Names: ACUVUE® OASYS™
  Arms: ACUVUE OASYS
Device: Lotrafilcon B contact lens (AIR OPTIX AQUA) — Silicone hydrogel contact lens worn for two weeks on a daily wear basis and cleaned nightly with one of three contact lens care solutions. The order of solutions was randomized, and a fresh pair of lenses was dispensed with each solution.
  Other Names: AIR OPTIX® AQUA
  Arms: AIR OPTIX AQUA
Device: Comfilcon A contact lens (Biofinity) — Silicone hydrogel contact lens worn for two weeks on a daily wear basis and cleaned nightly with one of three contact lens care solutions. The order of solutions was randomized, and a fresh pair of lenses was dispensed with each solution.
  Other Names: Biofinity®
  Arms: Biofinity

SUMMARY:
The purpose of this study was to evaluate the clinical performance of three differing contact lens care solutions when used in conjunction with three contact lenses.

DETAILED DESCRIPTION:
This study was conducted as three separate studies based on the contact lens brand dispensed. In each study, the contact lens was evaluated in conjunction with three solutions: Opti-Free Replenish, ReNu MultiPlus, and Clear Care. The total enrollment number of 75 represents a combined enrollment of the three studies, with some subjects participating in more than one study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Adapted contact lens wearer for at least one month.
* Spherical prescription range between +6.00 to -8.00 diopters.
* Astigmatism of less than or equal to 1.00 diopter in at least one eye.
* Normal eyes with no evidence of abnormality or disease.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Rigid Gas Permeable (RGP) contact lens wear in last 30 days.
* Concurrent ocular medication, systemic illness, or medical treatment that will affect ocular physiology, lens performance, or vision.
* Corneal infiltrates, scarring, or neovascularization within central 4 millimeters of cornea.
* Eye injury or surgery within 8 weeks prior to study.
* Aphakia, amblyopia, abnormal lacrimal secretions, ocular irritation, keratoconus, corneal irregularity, pregnancy, lactating, planning to become pregnant during the study, and participation in a concurrent clinical trial.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Modulus | 2 weeks
  Modulus is a measure of the stiffness of a contact lens material. Modulus is determined from the slope of the stress-strain curve created during tensile tests conducted on a sample of the material. Modulus is measured in mega Pascals (MPa). A higher modulus indicates a stiffer contact lens.
Bulbar hyperemia | 2 weeks
  Bulbar hyperemia is the injection (or redness) of the blood vessels in the tissues overlaying the white of the eye. Bulbar hyperemia is measured on a 0-4 scale, with 0=none, 1=trace, 2=mild, 3=moderate, and 4=severe. Half-grades are allowed.
Corneal staining type | 2 weeks
  An ophthalmic dye is used to highlight dead or degenerated corneal epithelial cells. The type of staining is measured over the five sectors of the cornea on a 0-4 scale, where 0=none, 1=micropunctate, 2=macropunctate, 3=coalesced macropunctate, and 4=patch (1mm). The five sectors are averaged to give a single score.
Upper palpebral roughness | 2 weeks
  The roughness of the inner lining of the upper eyelid is measured on a 0-4 scale, where 0=uniform appearance, 1=trace, 2=mild, 3=moderate, and 4=severe. Half grades are allowed.
High contrast visual acuity | 2 weeks
  High contrast visual acuity is a measure of the clearness of vision with full room illumination. Visual acuity is measured with a computer-generated, high contrast logMAR (logarithm minimum angle of resolution) chart.
End of day comfort | 2 weeks
  As assessed by the subject as a measure of the comfort of the contact lenses at the end of an average day. End of day comfort is recorded on an 11-point scale where 0=poor and 10=excellent.

CONTACTS AND LOCATIONS:
Locations (1):
- Visioncare Research Ltd., Farnham, Surrey, United Kingdom

REFERENCES:
- [Result] Program No 105358. Hall LA, Garofalo R, Young G. Clinical comparison of three contact lens systems in conjunction with senofilcon A, lotrafilcon B and comfilcon A daily wear lenses. American Academy of Optometry 2010.